CLINICAL TRIAL: NCT02348632
Title: A Long-Term Safety and Maintenance of Efficacy Study ofJZP-110 [(R)-2-amino-3 Phenylpropylcarbamate Hydrochloride] in the Treatment of Excessive Sleepiness in Subjects With Narcolepsy or Obstructive Sleep Apnea
Brief Title: "A Long-Term Safety Study of JZP-110 in the Treatment of Excessive Sleepiness in Subjects With Narcolepsy or OSA"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-005
Record Dates: First submitted 2015-01-15; First posted 2015-01-28 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Narcolepsy; Obstructive Sleep Apnea
MeSH Terms: conditions — Narcolepsy; Sleep Apnea, Obstructive | interventions — solriamfetol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 75 mg - 300 mg of JZP-110 (Other): Once Daily Dosing
  Interventions: Drug: JZP-110

INTERVENTIONS:
Drug: JZP-110

SUMMARY:
This is a Phase 3 study to assess the long-term safety and maintenance of efficacy of JZP-110 in subjects who have completed Study 14-002, 14-003, 14-004, 15-004, 15-005, ADX-N05 201, or ADX-N05 202.

ELIGIBILITY:
Major Inclusion Criteria:

1. Subject meets one of the following:

   1. Completed Study 14-002 or 14-003 (Group A)
   2. Completed Study 14-004, 15-004, 15-005, ADX-N05 201 or ADX-N05 202 (Group B)
2. Body mass index from 18 to <45 kg/m2
3. Consent to use a medically acceptable method of contraception
4. Willing and able to provide written informed consent

Major Exclusion Criteria:

1. Female subjects who are pregnant, nursing, or lactating
2. Any other clinically relevant medical, behavioral, or psychiatric disorder other than narcolepsy or OSA that is associated with excessive sleepiness
3. History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to DSM-5 criteria
4. Presence of any acutely unstable medical condition, behavioral or psychiatric disorder (including active suicidal ideation), or surgical history that could affect the safety of the subject or interfere with study efficacy or safety assessments, or the ability of the subject to complete the trial per the judgment of the Investigator
5. History of bariatric surgery within the past year or a history of roux-en-y procedure
6. Presence or history of significant cardiovascular disease
7. Use of any over the counter (OTC) or prescription medications that could affect the evaluation of excessive sleepiness
8. Received an investigational drug other than JZP-110 in the past 30 days or five half-lives (whichever is longer)
9. History of phenylketonuria (PKU) or history of hypersensitivity to phenylalanine-derived products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2015-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (80):
- United States (63):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Pulmonary Associates, Glendale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - UC San Diego Medical Center, La Jolla, California
  - So Cal Institute For Respiratory Diseases, Inc., Los Angeles, California
  - Pacific Sleep Medicine, Oceanside, California
  - The Research Center of Southern California, Oceanside, California
  - Stanford University Center for Narcolepsy, Redwood City, California
  - Pacific Research Network Inc., San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Critical care Pulmonary & Sleep Associates, LLC, Lakewood, Colorado
  - MD Clinical, Hallandale, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - Florida Pediatric Research Institute, Winter Park, Florida
  - Emory Sleep Center, Atlanta, Georgia
  - NeuroTrials Research Inc., Atlanta, Georgia
  - SleepMed of Central Georgia, Macon, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Illinois at Chicago Nursing School, Chicago, Illinois
  - Rowe Neurology Institute RNI - Lenexa, Lenexa, Kansas
  - Veritas Clinical Specialties LTD, Topeka, Kansas
  - Kentucky Research Group, Louisville, Kentucky
  - Advanced Neurodiagnostic Center, Metairie, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Neurocare, Inc., Newton, Massachusetts
  - Henry Ford Hospital Sleep Disorders & Research Center, Detroit, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - Minnesota Lung Center, Edina, Minnesota
  - Sleep Medicine & Research center, St. Lukes Hospital, Chesterfield, Missouri
  - University of Missouri, Columbia, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Clinilabs, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hickory Research Center, Hickory, North Carolina
  - Hickory Research Center, ARSM Research, LLC, Huntersville, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Northcoast Clinical Trials Inc., Beachwood, Ohio
  - Sleep Management Institute, Cincinnati, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Southwest Cleveland Sleep Research Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Sleep Medicine & Neuroscience Institute, Dublin, Ohio
  - Mercy St. Anne & Mercy St. Charles Sleep Disorders Center, Toledo, Ohio
  - Center for Sleep and Circadian Neurobiology, Philadelphia, Pennsylvania
  - UPMC Sleep Medicine Center, Pittsburgh, Pennsylvania
  - Lowcountry Lung Critical Care, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Sleep Med of South Carolina Clinical Research Solutions, Columbia, South Carolina
  - FutureSearch Trials of Neurology LP, Austin, Texas
  - Todd J. Swick, Houston, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - EVMS Sleep Medicine, Norfolk, Virginia
  - American Sleep Medicine, Vienna, Virginia
  - Swedish Medical Center, Seattle, Washington
- Canada (6):
  - London Health Sciences Centre, London, Ontario
  - Niagra Clinical Research, Niagra Falls, Ontario
  - Toronto Sleep Institute, Toronto, Ontario
  - Toronto Psychiatric Research Foundation, Toronto, Ontario
  - Pediatric Sleep Research Inc, Toronto, Ontario
  - CARSM Sleep Laboratory & Clinic, Montreal, Quebec
- Finland (2):
  - Unesta Research Center, Tampere
  - University of Turku , Sleep Research Centre, Turku
- France (6):
  - CHU de Dijon, Dijon
  - Grenoble University Hospital, La Tronche
  - Hospital Roger Salengro, Lille
  - Universite Paris 5 Hôtel-Dieu, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - CHU de Poitiers, Poitiers
- Germany (2):
  - Somnolab Dortmund, Dortmund
  - Klinische Forschung Schwerin GmbH, Schwerin
- Sleep Wake Center SEIN Heemstede, Heemstede, North Holland, Netherlands

REFERENCES:
- [Derived] Malhotra A, Strollo PJ Jr, Pepin JL, Schweitzer P, Lammers GJ, Hedner J, Redline S, Chen D, Chandler P, Bujanover S, Strohl K. Effects of solriamfetol treatment on body weight in participants with obstructive sleep apnea or narcolepsy. Sleep Med. 2022 Dec;100:165-173. doi: 10.1016/j.sleep.2022.08.005. Epub 2022 Aug 14. PMID 36084494
- [Derived] Weaver TE, Pepin JL, Schwab R, Shapiro C, Hedner J, Ahmed M, Foldvary-Schaefer N, Strollo PJ, Mayer G, Sarmiento K, Baladi M, Bron M, Chandler P, Lee L, Malhotra A. Long-term effects of solriamfetol on quality of life and work productivity in participants with excessive daytime sleepiness associated with narcolepsy or obstructive sleep apnea. J Clin Sleep Med. 2021 Oct 1;17(10):1995-2007. doi: 10.5664/jcsm.9384. PMID 34606437
- [Derived] Schweitzer PK, Strohl KP, Mayer G, Rosenberg R, Chandler P, Baladi M, Lee L, Malhotra A. Effects of solriamfetol in a long-term trial of participants with obstructive sleep apnea who are adherent or nonadherent to airway therapy. J Clin Sleep Med. 2021 Apr 1;17(4):659-668. doi: 10.5664/jcsm.8992. PMID 33179591
- [Derived] Malhotra A, Shapiro C, Pepin JL, Hedner J, Ahmed M, Foldvary-Schaefer N, Strollo PJ, Mayer G, Sarmiento K, Baladi M, Chandler P, Lee L, Schwab R. Long-term study of the safety and maintenance of efficacy of solriamfetol (JZP-110) in the treatment of excessive sleepiness in participants with narcolepsy or obstructive sleep apnea. Sleep. 2020 Feb 13;43(2):zsz220. doi: 10.1093/sleep/zsz220. PMID 31691827

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 645 subjects were enrolled in the study; 2 subjects withdrew from the study prior to receiving study drug. A total of 643 subjects received at least 1 dose of JZP-110 in the open-label phase and were included in the Safety Population.
Groups:
- JZP-110: Subjects completed a 2-week Titration phase. They then entered the maintenance phase of up to 50 weeks at the stable dose that was reached at the end of the Titration Phase.
- Placebo: Placebo administered orally, QD, for the 2-week randomized withdrawal period.
Period: Open-label Period
Arm/Group | JZP-110 | Placebo
Started | 643 | 0
Completed | 458 | 0
Not Completed | 185 | 0
Period: Randomized Withdrawal Period
Arm/Group | JZP-110 | Placebo
Started | 140 | 142
Completed | 137 | 141
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Open-label Period: 643 subjects comprised the safety population.
Arm/Group | Open-label Period
Number analyzed (Participants) | 643
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.31 (14.155)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 306
  Male | 337
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 109
  White | 506
  More than one race | 8
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Epworth Sleepiness Scale (ESS) Score
Description: Change in Epworth Sleepiness Scale (ESS) score during the 2-week randomized withdrawal period. The beginning of the randomized withdrawal period represents efficacy baseline. A negative change from baseline represents improvement in excessive sleepiness.
  The ESS is a self-administered questionnaire with 8 questions. Each activity is scored on a scale ranging from 0-3, with 0 = would never fall asleep, and 3 = high chance of falling asleep. The total score ranges from 0-24, with a higher number representing an increased propensity for sleepiness. An analysis of covariance (ANCOVA) was used for the analysis of ESS scores. This analysis included treatment group and randomization stratification factor (narcolepsy vs. OSA) as fixed effects. The ESS score at the beginning of the randomized withdrawal period was used as the covariate. The response variable was the change in ESS score from the beginning to the end of 2- week randomized withdrawal period.
Time Frame: Start of randomized withdrawal phase to end of randomized withdrawal (2 weeks)
Population: 282 subjects were randomized into the randomized withdrawal period. Two subjects who were treated in the randomized withdrawal period did not have evaluable efficacy data during that period. Therefore, the mITT Population comprised 280 subjects, 141 who received placebo and 139 who received JZP-110.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Groups:
- Placebo: JZP-110 administered orally, QD, for the 2-week randomized withdrawal period, at the same dose subjects were currently receiving.
Arm/Group | JZP-110 | Placebo
Number analyzed (Participants) | 139 | 141
points on a scale | 1.6 (0.41) | 5.3 (0.41)

2. Secondary Outcome: Subjects Reported as Worse on the Patient Global Impression of Change (PGIc)
Description: Percentage of subjects reported as worse (minimally worse, much worse, or very much worse) on the PGIc during the 2-week randomized withdrawal period. The beginning of the randomized withdrawal period represents efficacy baseline.
Time Frame: Beginning of randomized withdrawal phase to end of the randomized withdrawal phase (2 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | JZP-110 | Placebo
Number analyzed (Participants) | 139 | 141
percentage of subjects | 28.2 | 64.5

3. Secondary Outcome: Subjects Reported as Worse on the Clinical Global Impression of Change (CGIc)
Description: Subjects reported as worse (very much worse, much worse, and minimally worse) on the CGIc during the 2-week randomized withdrawal period. The beginning of the randomized withdrawal period represents efficacy baseline.
Time Frame: Beginning of randomized withdrawal phase to end of the randomized withdrawal phase (2 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | JZP-110 | Placebo
Number analyzed (Participants) | 139 | 141
percentage of subjects | 28.7 | 63.8

ADVERSE EVENTS:
Time Frame: The Safety Population consisted of all subjects who received at least 1 dose of study medication. Adverse events are reported across the entire study (e.g., the open-label and randomized withdrawal periods combined).
Arm/Group | JZP-110 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/643 | 0/142
Serious Adverse Events (participants affected / at risk) | 27/643 | 0/142
Other Adverse Events (participants affected / at risk) | 269/643 | 3/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JZP-110 (N=643) | Placebo (N=142)
Deep vein thrombosis (Vascular disorders) | 1 | 0
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | NA
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Agitation (Psychiatric disorders) | 2 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0
Ear canal injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 1 | 0
Cluster headache (Nervous system disorders) | 2 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Ear and labyrinth disorders) | 2 | 0
Duodenal ulcer haemorrhage (Ear and labyrinth disorders) | 1 | 0
Gastrointestinal inflammation (Ear and labyrinth disorders) | 1 | 0
Nausea (Ear and labyrinth disorders) | 1 | 0
Vomiting (Ear and labyrinth disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JZP-110 (N=643) | Placebo (N=142)
Headache (Nervous system disorders) | 71 | 0
Anxiety (Psychiatric disorders) | 46 | 0
Insomnia (Psychiatric disorders) | 51 | 1
Nausea (Gastrointestinal disorders) | 57 | 1
Dry mouth (Gastrointestinal disorders) | 47 | 0
Decreased appetite (Metabolism and nutrition disorders) | 32 | 0
Nasopharyngitis (Infections and infestations) | 54 | 1
Upper respiratory tract infection (Infections and infestations) | 32 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT02348632/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT02348632/SAP_001.pdf